CLINICAL TRIAL: NCT04262531
Title: Body Composition and Clinical Outcomes in Critically Ill Patients: A Prospective Observational Study
Brief Title: Body Composition Study in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Other Study IDs: MREC ID NO: 2019615-7520
Record Dates: First submitted 2020-01-15; First posted 2020-02-10 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Critical Illness; Muscle Loss
Keywords: Critical Illness; muscle; mortality
MeSH Terms: conditions — Critical Illness; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center prospective observational study that aimed to describe the trajectory of change in body composition among critically ill patients who were able to function independently prior to admission. Ultrasound measurement of the quadriceps muscle and bioelectrical impedance analysis will be conducted at baseline, day 7, day 14 and before ICU discharge. The relationship between the change of body composition and clinical outcomes, activities of daily living and quality of life at 6-month post ICU admission will be investigated. Further, the association between nutritional (energy and protein) intake and change in body composition will also be investigated.

DETAILED DESCRIPTION:
Malnutrition is associated with poor clinical outcomes. Nutritional status is closely linked with body lean mass, specifically the skeletal muscle. Several tool s had been suggested to determine nutrition risk and status for critically ill patients such as The Nutrition Risk in Critically Ill (NUTRIC) and subjective global assessment (SGA). However, they are surrogate (NUTRIC) or subjective (SGA) measures of nutritional status. Ideally, clinicians should measure muscle directly to determine the patient nutritional status. Several imaging techniques allow direct and accurate measurement of muscle mass, these include magnetic resonance imaging (MRI) and computed-tomography (CT). However, the measurement of MRI and CT involves the transfer of patients out of the intensive care unit or expose the patient to radiation (CT) and therefore it is not justifiable to conduct MRI or CT for the sole purpose of measuring body composition. Ultrasound and bioelectrical impedance analysis (BIA) are non-invasive and can be conducted at the bedside and therefore are promising techniques in assessing patients' nutritional status. Ultrasound measurement of quadriceps thickness and rectus femoris cross-sectional area can measure muscle directly and are widely used in the research setting. BIA phase angle is a direct measure of cell integrity and is an independent predictor of mortality in the ICU.

This study aimed to describe the trajectory of change in body composition and investigate the relationship of the changes with clinical outcomes and activities of daily living and quality of life at 6-month post ICU admission. Further, the association between nutritional (energy and protein) intake and change in body composition will also be investigated to determine if the ultrasound or BIA measurements of body composition can help to assess the response to nutritional intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Mechanically ventilated* within 48 hours of ICU admission
* Expected to stay in the ICU ≥96 hours
* CT imaging is done within 72 hours prior and after ICU admission (only applicable for CT analysis)

Exclusion Criteria:

* Pregnant
* Expected death or discussion to withdraw life-sustaining treatments within this hospitalization
* Patients in the hospital (either in the ward or ICU) ≥5 days in the past 2 weeks before enrolment
* Not ambulating independently prior to illness that led to ICU admission (use of gait aid permitted). Also exclude if unable to walk 50 feet (15 meters) prior to hospitalization
* Pre-existing (chronic or acute presentation) primary systemic neuromuscular disease (e.g. Guillain Barre)
* Patient on pacemaker
* Bilateral lower limb deep vein thrombosis
* Presence of iliopsoas abscess or hematoma (only applicable for CT analysis)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult mechanically ventilated critically ill patients who are expected to stay at least 96 hours in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Rectus Femoris Thickness | Change in rectus femoris thickness and cross-sectional area at day 7, 14 and within 72 hours of ICU discharge compared with baseline (Day 1 of ICU admission)
  Change in rectus femoris thickness
Rectus Femoris Cross-sectional area | Change in rectus femoris thickness and cross-sectional area at day 7, 14 and within 72 hours of ICU discharge compared with baseline (Day 1 of ICU admission)
  Change in rectus femoris cross-sectional area

SECONDARY OUTCOMES:
Ultrasound quadriceps echogenicity | Change in quadriceps echogenicity, pennation angle and fascicle length at day 7, 14 and within 72 hours of ICU discharge compared with baseline (Day 1 of ICU admission)
  Change in quadriceps echogenicity
Ultrasound quadriceps pennation angle | Change in quadriceps echogenicity, pennation angle and fascicle length at day 7, 14 and within 72 hours of ICU discharge compared with baseline (Day 1 of ICU admission)
  Change in quadriceps pennation angle
Ultrasound quadriceps fascicle length | Change in quadriceps echogenicity, pennation angle and fascicle length at day 7, 14 and within 72 hours of ICU discharge compared with baseline (Day 1 of ICU admission)
  Change in quadriceps fascicle length
Bioelectrical Impedance Analysis (BIA) phase angle | Change in whole body BIA phase angle at day 7, 14 and within 72 hours of ICU discharge compared with baseline (Day 1 of ICU admission)
  Change in whole body BIA phase angle

OTHER OUTCOMES:
Percentage of participant who died (Mortality) | Mortality at day 28 and day 60 (calculated from the first day of ICU admission)
  Mortality at day 28, day 60, in the ICU and in the Hospital
Survivors' long-term quality of life status | 6 months after ICU admission
  Survivors' quality of life status at 6 months of ICU admission by administering Euro Quality of Life 5-level questionnaire (EQ-5D-5L) via telephone interview. The are 5 questions and each question will have 5 categories (Level 1 is the best and level 5 is worst).
Katz Activities of Daily Living (ADL) | 6 months after ICU admission
  Survivors' ADL status at 6 months of ICU admission by administering Katz ADL questionnaire via telephone interview. Katz ADL has 5 questions with score ranging from 0 to 6, higher score is better.
Lawton Instrumental Activities of Daily Living (IADL) | 6 months after ICU admission
  Survivors' IADL status at 6 months of ICU admission by administering Lawton IADL questionnaire via telephone interview. Lawton IADL has 8 questions with score ranging from 0 to 8, the higher score is better.

CONTACTS AND LOCATIONS:
Overall Officials: Ng Ching Choe Chloe, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Lew CCH, Yandell R, Fraser RJL, Chua AP, Chong MFF, Miller M. Association Between Malnutrition and Clinical Outcomes in the Intensive Care Unit: A Systematic Review [Formula: see text]. JPEN J Parenter Enteral Nutr. 2017 Jul;41(5):744-758. doi: 10.1177/0148607115625638. Epub 2016 Feb 2. PMID 26838530
- [Background] Lee ZY, Heyland DK. Determination of Nutrition Risk and Status in Critically Ill Patients: What Are Our Considerations? Nutr Clin Pract. 2019 Feb;34(1):96-111. doi: 10.1002/ncp.10214. Epub 2018 Nov 23. PMID 30468264
- [Background] White JV, Guenter P, Jensen G, Malone A, Schofield M; Academy Malnutrition Work Group; A.S.P.E.N. Malnutrition Task Force; A.S.P.E.N. Board of Directors. Consensus statement: Academy of Nutrition and Dietetics and American Society for Parenteral and Enteral Nutrition: characteristics recommended for the identification and documentation of adult malnutrition (undernutrition). JPEN J Parenter Enteral Nutr. 2012 May;36(3):275-83. doi: 10.1177/0148607112440285. PMID 22535923
- [Background] Prado CM, Heymsfield SB. Lean tissue imaging: a new era for nutritional assessment and intervention. JPEN J Parenter Enteral Nutr. 2014 Nov;38(8):940-53. doi: 10.1177/0148607114550189. Epub 2014 Sep 19. PMID 25239112
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Mourtzakis M, Parry S, Connolly B, Puthucheary Z. Skeletal Muscle Ultrasound in Critical Care: A Tool in Need of Translation. Ann Am Thorac Soc. 2017 Oct;14(10):1495-1503. doi: 10.1513/AnnalsATS.201612-967PS. PMID 28820608
- [Background] Thibault R, Makhlouf AM, Mulliez A, Cristina Gonzalez M, Kekstas G, Kozjek NR, Preiser JC, Rozalen IC, Dadet S, Krznaric Z, Kupczyk K, Tamion F, Cano N, Pichard C; Phase Angle Project Investigators. Fat-free mass at admission predicts 28-day mortality in intensive care unit patients: the international prospective observational study Phase Angle Project. Intensive Care Med. 2016 Sep;42(9):1445-53. doi: 10.1007/s00134-016-4468-3. Epub 2016 Aug 11. PMID 27515162
- [Background] Lee ZY, Ong SP, Ng CC, Yap CSL, Engkasan JP, Barakatun-Nisak MY, Heyland DK, Hasan MS. Association between ultrasound quadriceps muscle status with premorbid functional status and 60-day mortality in mechanically ventilated critically ill patient: A single-center prospective observational study. Clin Nutr. 2021 Mar;40(3):1338-1347. doi: 10.1016/j.clnu.2020.08.022. Epub 2020 Aug 28. PMID 32919818